CLINICAL TRIAL: NCT02073747
Title: The Various Effects of Gaseous Albuterol on Serum Lactate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center of Southern Nevada (Other)
Responsible Party: Principal Investigator, Joseph Anthony Zitek, MD, University Medical Center of Southern Nevada
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: EM 2014.01
Record Dates: First submitted 2014-02-19; First posted 2014-02-27 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Asthma
Keywords: Albuterol; Serum Lactate; Lactic Acidosis; Asthma
MeSH Terms: conditions — Asthma; Acidosis, Lactic | interventions — Saline Solution; Sodium Chloride; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline Control Group (Placebo Comparator): Control group will be administered a one hour normal saline inhaled treatment.
  Interventions: Drug: Normal Saline
- Albuterol Trial Group (Active Comparator): Trial group to be administered one hour treatment of ten milligrams of inhaled albuterol
  Interventions: Drug: Albuterol

INTERVENTIONS:
Drug: Normal Saline — One hour inhaled normal saline
  Other Names: NS; Saline
  Arms: Normal Saline Control Group
Drug: Albuterol — One hour inhaled ten milligrams of albuterol
  Other Names: Ventilin; Proventil
  Arms: Albuterol Trial Group

SUMMARY:
Empirical data from physician observation indicates an increase in serum lactate in acute asthmatic patients being treated with inhaled albuterol therapy.

It is not clear if this increased serum lactate is in response to a physiological response to the asthmatic process or from the albuterol treatment.

This study is designed to determine if administration of inhaled albuterol increases serum lactate in healthy subjects.

DETAILED DESCRIPTION:
Approximately 30 healthy volunteers will be randomized to Albuterol or placebo. We powered our study to detect a difference of 0.5 mmol/L, but hypothesize that the difference will be greater than 1.0 mmol/L.

All volunteer subjects will sign a written consent, approved by the Institutional Review Board. The intended pool of volunteers will be from residents, attendings, and medical students in the hospital. The consent form will clearly specify that their participation in the study will not impact their academic status or employment.

The subjects randomized to the Albuterol arm will receive a one hour 10 mg continuous Albuterol nebulizer treatment. Those randomized to placebo will receive a one-hour saline nebulizer treatment. The chief pharmacist for the study will randomly assign a number between one and thirty to fifteen Albuterol treatments and fifteen placebo treatments.

Subjects will be monitored with cardiac monitor and serum lactate levels will be drawn every 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older

Exclusion Criteria:

* Pregnant
* Prisoner
* beta agonist allergy
* hypokalemia
* taking furosemide, insulin, thiazide diuretics, metformin or acetazolamide
* coronary artery disease
* hyperthyroidism
* abnormal heart rhythm
* baseline serum lactate level >2.2 mmol/L
* baseline heart rate > 120

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Zitek, MD, Principal Investigator — Emergency Medicine Residency Faculty
Locations (1):
- University Medical Center of Southern Nevada, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Background] Appel D, Rubenstein R, Schrager K, Williams MH Jr. Lactic acidosis in severe asthma. Am J Med. 1983 Oct;75(4):580-4. doi: 10.1016/0002-9343(83)90436-9. PMID 6414303
- [Background] Roncoroni AJ, Adrougue HJ, De Obrutsky CW, Marchisio ML, Herrera MR. Metabolic acidosis in status asthmaticus. Respiration. 1976;33(2):85-94. doi: 10.1159/000193721. PMID 778959
- [Background] Manthous CA. Lactic acidosis in status asthmaticus : three cases and review of the literature. Chest. 2001 May;119(5):1599-602. doi: 10.1378/chest.119.5.1599. PMID 11348975
- [Background] Maury E, Ioos V, Lepecq B, Guidet B, Offenstadt G. A paradoxical effect of bronchodilators. Chest. 1997 Jun;111(6):1766-7. doi: 10.1378/chest.111.6.1766. PMID 9187208
- [Background] Chaulier K, Chalumeau S, Ber CE, Bret M, Rimmele T. [Metabolic acidosis in a context of acute severe asthma]. Ann Fr Anesth Reanim. 2007 Apr;26(4):352-5. doi: 10.1016/j.annfar.2007.01.016. Epub 2007 Mar 8. French. PMID 17349773
- [Background] Rodrigo GJ, Rodrigo C. Elevated plasma lactate level associated with high dose inhaled albuterol therapy in acute severe asthma. Emerg Med J. 2005 Jun;22(6):404-8. doi: 10.1136/emj.2003.012039. PMID 15911945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were recruited from the investigators' friends and family.
Period: Overall Study
Arm/Group | Normal Saline Control Group | Albuterol Trial Group
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Albuterol: Study group
- Normal Saline: Control group
- Total: Total of all reporting groups
Arm/Group | Albuterol | Normal Saline | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [24.5 to 30] | 28 [26.3 to 34.5] | 28.5 [26 to 32.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 10 | 7 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Change From Baseline Serum Lactate Following a One Hour Albuterol Nebulizer Treatment.
Description: We powered our study to detect a difference of 0.5 mmol/L between pre and post-treatment lactate levels, but hypothesize that the difference will be greater than 1.0 mmol/L.
Time Frame: Change in serum lactate from baseline to 1 hour
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Normal Saline Control Group | Albuterol Trial Group
Number analyzed (Participants) | 14 | 14
mmol/L | -0.15 [-0.39 to 0.09] | 0.77 [0.52 to 1.02]

ADVERSE EVENTS:
Groups:
- Albuterol: Study group; 10 mg of nebulizer albuterol
Arm/Group | Albuterol | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No